CLINICAL TRIAL: NCT06242444
Title: A Randomized, Examiner Blind, Crossover, in Situ Erosion Study To Investigate The Efficacy Of An Experimental Dentifrice In Remineralization Of Softened Enamel Compared To Placebo and Reference Dentifrices
Brief Title: An Erosion Study to Investigate the Efficacy of an Experimental Dentifrice to Remineralize Enamel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 300057
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Dentifrice (Experimental): Participants will brush the buccal surfaces of their natural teeth using 1.5+/- 0.1 grams (g) of the experimental dentifrice containing 1150 ppm fluoride and 5 percent (%) potassium nitrate (KNO3) for 25 timed seconds and then swish the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. Participants will use the dentifrice under supervision of the study staff while the intraoral appliance is in place in Treatment Periods 1 to 3. There will be a washout period of a minimum of 3 days prior to each treatment during which the participants will use their own dentifrice for at least one day, and a 0 ppm fluoride washout dentifrice for two days.
  Interventions: Drug: Experimental Dentifrice
- Placebo Control Dentifrice (Placebo Comparator): Participants will brush the buccal surfaces of their natural teeth using 1.5+/- 0.1 g of the placebo dentifrice containing 0 ppm fluoride and 5% KNO3 for 25 timed seconds and then swish the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. Participants will use the dentifrice under supervision of the study staff while the intraoral appliance is in place in Treatment Periods 1 to 3. There will be a washout period of a minimum of 3 days prior to each treatment during which the participants will use their own dentifrice for at least one day, and a 0 ppm fluoride washout dentifrice for two days.
  Interventions: Drug: Placebo Control Dentifrice
- Reference Dentifrice (Active Comparator): Participants will brush the buccal surfaces of their natural teeth using 1.5+/- 0.1 g of the reference dentifrice containing 1100 ppm fluoride as stannous fluoride (SnF2) for 25 timed seconds and then swish the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. Participants will use the dentifrice under supervision of the study staff while the intraoral appliance is in place in Treatment Periods 1 to 3. There will be a washout period of a minimum of 3 days prior to each treatment during which the participants will use their own dentifrice for at least one day, and a 0 ppm fluoride washout dentifrice for two days.
  Interventions: Drug: Reference Dentifrice

INTERVENTIONS:
Drug: Experimental Dentifrice — Dentifrice containing 1150 ppm fluoride and 5% KNO3.
  Arms: Experimental Dentifrice
Drug: Placebo Control Dentifrice — Dentifrice containing 0 ppm fluoride and 5% KNO3.
  Arms: Placebo Control Dentifrice
Drug: Reference Dentifrice — Dentifrice containing 1100 ppm fluoride as SnF2.
  Other Names: Crest Pro-Health Densify Daily Protection
  Arms: Reference Dentifrice

SUMMARY:
The purpose of this study is to investigate the ability of an experimental dentifrice containing 1150 parts per million (ppm) fluoride to remineralize acid-softened dental enamel and help prevent further demineralization compared to a 0 ppm fluoride placebo dentifrice and a marketed, fluoride-containing dentifrice (Reference Dentifrice).

DETAILED DESCRIPTION:
This will be a randomized, controlled, single center, single-blind, 3 period, 3 treatment, cross-over, in situ design study. Previously demineralized bovine enamel specimens will be placed intra orally using a palatal appliance and the remineralizing performance of the experimental, reference and placebo dentifrices will be evaluated at 4 and 12 hours post toothbrushing, based on surface micro hardness measurements of the bovine enamel specimens. At each treatment visit, once the palatal the appliance is fitted in the mouth, a five minute equilibration period will ensue following which each participant will brush their teeth with their assigned product. Participants will remove the appliance for 30 minutes at 4 and 8.5 hours post brushing and will remove and store the appliance 13 hours post brushing (12 hours intraoral exposure). Sufficient participants will be screened to randomize approximately 33 participants to study treatment to ensure approximately 30 participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is between the ages of 18-65 years, inclusive.
* Participant is willing and able to comply with scheduled visits, and other study procedures and restrictions.
* Participant is in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant with generally good oral health that fulfil all of the following:

  1. Having an unstimulated salivary flow rate of at least 0.2 milliliter per minute (mL/minute) and a stimulated salivary flow rate of at least 0.8 mL/minute.
  2. Having a maxillary dental arch suitable for the retention of the palatal appliance.
  3. Having no lesions of the oral cavity that could interfere with the study evaluations.

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family (employees of the study site and associated academic institutes who are not directly involved in the conduct of the study are eligible to be considered as participants.)
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study or who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who, in the opinion of the investigator or medically qualified designee, can't comply with study requirements or who should not participate in the study for other reasons.
* Participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* Participant taking medication that may interfere significantly with the saliva flow in the judgment of the investigator. Should new medications that may interfere with the saliva flow be added, a second salivary flow test will be performed.
* Participant with any condition that would impact on their safety or wellbeing or affect their ability to understand and follow study procedures and requirements.
* Participant with any sign of grossly carious lesions (active), moderate or severe periodontal conditions, or severe tooth wear. Participant presenting at screening with minor caries may continue in the study if their carious lesions are repaired prior to the first treatment visit of the study.
* Participant who wears an oral piercing or oral appliance or orthodontia (besides participants wearing permanent lower retainers, which are eligible).
* Participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 34 participants were screened of which 33 participants were randomized as per crossover design to receive either one of the 6 treatment sequences: Sequence ABC, Sequence ACB, Sequence BAC, Sequence BCA, Sequence CAB, Sequence CBA where Treatment A=Test Dentifrice, Treatment B=Placebo Control Dentifrice, Treatment C=Reference Dentifrice. All 33 randomized participants completed the study.
Groups:
- Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 grams (g) of the Test Dentifrice containing 1150 parts per million (ppm) fluoride and 5 percent (%) potassium nitrate (KNO3) once on Day 1 of Treatment Period 1 (Treatment A) followed by 1.5+/-0.1 g of Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 2 (Treatment B) and further followed by 1.5+/-0.1 g of Reference Dentifrice containing 1100 ppm fluoride as stannous fluoride (SnF2) once on Day 1 of Treatment Period 3 (Treatment C). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
- Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of the Test Dentifrice containing 1150 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 1 (Treatment A) followed by 1.5+/-0.1 g of Reference Dentifrice containing 1100 ppm fluoride as SnF2 once on Day 1 of Treatment Period 2 (Treatment C) and further followed by 1.5+/-0.1 g of Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 3 (Treatment B). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
- Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 1 (Treatment B) followed by 1.5+/-0.1 g of the Test Dentifrice containing 1150 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 2 (Treatment A) and further followed by 1.5+/-0.1 g of Reference Dentifrice containing 1100 ppm fluoride as SnF2 once on Day 1 of Treatment Period 3 (Treatment C). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
- Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 1 (Treatment B) followed by 1.5+/-0.1 g of the Reference Dentifrice containing 1100 ppm fluoride as SnF2 once on Day 1 of Treatment Period 2 (Treatment C) and further followed by 1.5+/-0.1 g of Test Dentifrice containing 1150 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 3 (Treatment A). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
- Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of Reference Dentifrice containing 1100 ppm fluoride as SnF2 once on Day 1 of Treatment Period 1 (Treatment C) followed by 1.5+/-0.1 g of the Test Dentifrice containing 1150 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 2 (Treatment A) and further followed by 1.5+/-0.1 g of Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 3 (Treatment B). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
- Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice): Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of Reference Dentifrice containing 1100 ppm fluoride as SnF2 once on Day 1 of Treatment Period 1 (Treatment C) followed by 1.5+/-0.1 g of the Placebo Control Dentifrice containing 0 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 2 (Treatment B) and further followed by 1.5+/-0.1 g of Test Dentifrice containing 1150 ppm fluoride and 5% KNO3 once on Day 1 of Treatment Period 3 (Treatment A). Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds. There was a washout period of a minimum of 3 days prior to each treatment.
Period: Treatment Period 1 (2 Days)
Arm/Group | Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice) | Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice) | Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice) | Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice) | Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice) | Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice)
Started | 5 | 5 | 6 | 6 | 5 | 6
Completed | 5 | 5 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (3 Days)
Arm/Group | Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice) | Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice) | Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice) | Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice) | Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice) | Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice)
Started | 5 | 5 | 6 | 6 | 5 | 6
Completed | 5 | 5 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (2 Days)
Arm/Group | Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice) | Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice) | Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice) | Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice) | Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice) | Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice)
Started | 5 | 5 | 6 | 6 | 5 | 6
Completed | 5 | 5 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (3 Days)
Arm/Group | Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice) | Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice) | Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice) | Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice) | Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice) | Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice)
Started | 5 | 5 | 6 | 6 | 5 | 6
Completed | 5 | 5 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (2 Days)
Arm/Group | Sequence ABC (Test Dentifrice + Placebo Control Dentifrice + Reference Dentifrice) | Sequence ACB (Test Dentifrice + Reference Dentifrice + Placebo Control Dentifrice) | Sequence BAC (Placebo Control Dentifrice + Test Dentifrice + Reference Dentifrice) | Sequence BCA (Placebo Control Dentifrice + Reference Dentifrice + Test Dentifrice) | Sequence CAB (Reference Dentifrice + Test Dentifrice + Placebo Control Dentifrice) | Sequence CBA (Reference Dentifrice + Placebo Control Dentifrice + Test Dentifrice)
Started | 5 | 5 | 6 | 6 | 5 | 6
Completed | 5 | 5 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were randomized in the study.
Groups:
- Overall Study Participants: Participants brushed the buccal surfaces of their natural teeth using 1.5+/-0.1 g of the Test Dentifrice (Treatment A) containing 1150 ppm fluoride and 5% KNO3, Placebo Control Dentifrice (Treatment B) containing 0 ppm fluoride and 5% KNO3, Reference Dentifrice (Treatment C) containing 1100 ppm fluoride as SnF2 on Day 1 of Treatment Period 1, 2 or 3 as per randomization schedule. Participants used the assigned dentifrice under supervision of the study staff while the intraoral appliance was in place and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black or African American | 9
  White | 20

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Percent Surface Microhardness Recovery (%SMHR) at 4 Hours (Test Dentifrice Versus (vs.) Placebo Control Dentifrice)
Description: %SMHR was used to measure the ability of the dentifrice to remineralize enamel. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and the extent of remineralization was evaluated using surface microhardness (SMH) technique to yield the %SMHR. The enamel specimens were evaluated both prior to and after intra-oral exposure and indentation lengths were measured. The %SMHR was derived as [(E1-R)/(E1-B)] * 100 where: B = indentation length (micrometre [μm]) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 4 hours in situ remineralization.
Time Frame: At 4 hours of intra-oral exposure following treatment on Day 1 of each treatment period (each treatment period was of 2 days with 3 days washout in between)
Population: ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: percent SMHR
Groups:
- Test Dentifrice (Treatment A): Participants brushed the buccal surfaces of their natural teeth using 1.5+/- 0.1 g of the Test Dentifrice (Treatment A) containing 1150 ppm fluoride and 5% KNO3 for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds, once on Day 1 of Treatment Periods 1 to 3 as per randomization schedule. Participants used the dentifrice under supervision of the study staff while the intraoral appliance was in place.
- Placebo Control Dentifrice (Treatment B): Participants brushed the buccal surfaces of their natural teeth using 1.5+/- 0.1 g of the Placebo Control Dentifrice (Treatment B) containing 0 ppm fluoride and 5% KNO3 for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds, once on Day 1 of Treatment Periods 1 to 3 as per randomization schedule. Participants used the dentifrice under supervision of the study staff while the intraoral appliance was in place.
Arm/Group | Test Dentifrice (Treatment A) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
percent SMHR | 32.20 (2.021) | 23.85 (2.021)
Statistical Analysis 1: Comparison: Test Dentifrice (Treatment A) vs Placebo Control Dentifrice (Treatment B); Test type: Superiority; p = 0.0012, Mixed Models Analysis; Adjusted Mean Difference = 8.35, 95% CI 2-sided [3.42 to 13.28], Standard Error of Mean 2.465 — Adjusted mean difference was calculated as Test Dentifrice minus Placebo Control Dentifrice

2. Secondary Outcome: Adjusted Mean Percent Relative Erosion Resistance (%RER) at 4 Hours (Test Dentifrice vs. Placebo Control Dentifrice)
Description: %RER was used to measure the ability of the dentifrice to protect enamel from further acid-induced demineralization by both acid protection and remineralization. SMH technique was used to calculate %RER. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and further treated with acid ex situ followed by additional SMH evaluations to calculate %RER. The %RER was derived as [(E1-E2)/(E1-B)] * 100 where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), E2 = indentation length (μm) after second erosive challenge (with a commercially available grapefruit juice).
Time Frame: as for outcome 1
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent RER
Arm/Group | Test Dentifrice (Treatment A) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
percent RER | -11.56 (3.024) | -48.89 (3.024)
Statistical Analysis 1: Comparison: Test Dentifrice (Treatment A) vs Placebo Control Dentifrice (Treatment B); Test type: Superiority; p < .0001, Mixed Models Analysis; Adjusted Mean Difference = 37.33, 95% CI 2-sided [30.90 to 43.76], Standard Error of Mean 3.217 — Adjusted mean difference was calculated as Test Dentifrice minus Placebo Control Dentifrice

3. Secondary Outcome: Adjusted Mean %SMHR at 4 Hours (Test Dentifrice vs. Reference Dentifrice)
Description: %SMHR was used to measure the ability of the dentifrice to remineralize enamel. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and the extent of remineralization was evaluated using surface SMH technique to yield the %SMHR. The enamel specimens were evaluated both prior to and after intra-oral exposure and indentation lengths were measured. The %SMHR was derived as [(E1-R)/(E1-B)] * 100 where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 4 hours in situ remineralization.
Time Frame: as for outcome 1
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent SMHR
Groups:
- Reference Dentifrice (Treatment C): Participants brushed the buccal surfaces of their natural teeth using 1.5+/- 0.1 g of the Reference Dentifrice (Treatment C) containing 1100 ppm fluoride as SnF2 for 25 timed seconds and then swished the resulting dentifrice slurry around the mouth, without further brushing, for a timed period of 95 seconds, once on Day 1 of Treatment Periods 1 to 3 as per randomization schedule. Participants used the dentifrice under supervision of the study staff while the intraoral appliance was in place.
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C)
Number analyzed (Participants) | 33 | 33
percent SMHR | 32.20 (2.021) | 28.25 (2.019)
Statistical Analysis 1: Comparison: Test Dentifrice (Treatment A) vs Reference Dentifrice (Treatment C); Test type: Superiority; p = 0.1138, Mixed Models Analysis; Adjusted Mean Difference = 3.95, 95% CI 2-sided [-0.97 to 8.87], Standard Error of Mean 2.462 — Adjusted mean difference was calculated as Test Dentifrice minus Reference Dentifrice

4. Secondary Outcome: Adjusted Mean %SMHR at 12 Hours
Description: %SMHR was used to measure the ability of the dentifrice to remineralize enamel. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and the extent of remineralization was evaluated using SMH technique to yield the %SMHR. The enamel specimens were evaluated both prior to and after intra-oral exposure and indentation lengths were measured. The %SMHR was derived as [(E1-R)/(E1-B)] * 100 where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 12 hours in situ remineralization.
Time Frame: At 12 hours of intra-oral exposure following treatment on Day 1 of each treatment period (each treatment period was of 2 days with 3 days washout in between)
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent SMHR
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33 | 33
percent SMHR | 39.32 (1.826) | 36.66 (1.824) | 33.66 (1.826)

5. Secondary Outcome: Adjusted Mean %RER at 4 Hours (Test Dentifrice vs. Reference Dentifrice)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent RER
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C)
Number analyzed (Participants) | 33 | 33
percent RER | -11.56 (3.024) | -13.78 (3.022)
Statistical Analysis 1: Comparison: Test Dentifrice (Treatment A) vs Reference Dentifrice (Treatment C); Test type: Superiority; p = 0.4930, Mixed Models Analysis; Adjusted Mean Difference = 2.22, 95% CI 2-sided [-4.21 to 8.64], Standard Error of Mean 3.213 — Adjusted mean difference was calculated as Test Dentifrice minus Reference Dentifrice

6. Secondary Outcome: Adjusted Mean %RER at 12 Hours
Description: as for outcome 2
Time Frame: as for outcome 4
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent RER
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33 | 33
percent RER | -0.28 (2.760) | 0.19 (2.759) | -26.98 (2.760)

7. Secondary Outcome: Adjusted Mean Enamel Fluoride Uptake (EFU) at 4 and 12 Hours
Description: EFU is a measure of how much fluoride has been incorporated into the enamel during the process of remineralization. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and chemically analyzed to measure the amount of fluoride incorporated into the enamel by the dentifrice treatment.
Time Frame: At 4 and 12 hours of intra-oral exposure following treatment on Day 1 of each treatment period (each treatment period was of 2 days with 3 days washout in between)
Population: ITT population.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: microgram fluoride per square centimeter
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33 | 33
microgram fluoride per square centimeter
  At 4 hours of intra-oral exposure | 4.80 [4.31 to 5.35] | 3.81 [3.42 to 4.25] | 2.20 [1.98 to 2.45]
  At 12 hours of intra-oral exposure | 4.80 [4.41 to 5.22] | 3.89 [3.58 to 4.24] | 2.45 [2.25 to 2.66]

8. Secondary Outcome: Adjusted Mean Acid Resistance Ratio (ARR) at 4 and 12 Hours
Description: ARR was used to measure the resistance of the remineralized enamel to further acid softening. SMH technique was used to calculate ARR. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and further treated with acid ex situ followed by additional SMH evaluations to calculate ARR. The ARR was derived as 1 - [(E2-R)/(E1-B)] where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), E2 = indentation length (μm) after second erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 4 and 12 hours in situ remineralization.
Time Frame: as for outcome 7
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33 | 33
ratio
  At 4 hours of intra-oral exposure | 0.562 (0.0214) | 0.580 (0.0214) | 0.273 (0.0214)
  At 12 hours of intra-oral exposure | 0.604 (0.0200) | 0.635 (0.0200) | 0.394 (0.0200)

9. Secondary Outcome: Adjusted Mean %SMHR at 4 and 12 Hours (Reference Dentifrice vs Placebo Control Dentifrice)
Description: %SMHR was used to measure the ability of the dentifrice to remineralize enamel. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatment in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and the extent of remineralization was evaluated using SMH technique to yield the %SMHR. The enamel specimens were evaluated both prior to and after intra-oral exposure and indentation lengths were measured. The %SMHR was derived as [(E1-R)/(E1-B)] * 100 where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 4 and 12 hours in situ remineralization.
Time Frame: as for outcome 7
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent SMHR
Arm/Group | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
percent SMHR
  At 4 hours of intra-oral exposure | 28.25 (2.019) | 23.85 (2.021)
  At 12 hours of intra-oral exposure | 36.66 (1.824) | 33.66 (1.826)
Statistical Analysis 1: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 4 hours of intra-oral exposure; Test type: Superiority; p = 0.0789, Mixed Models Analysis; Adjusted Mean Difference = 4.40, 95% CI 2-sided [-0.52 to 9.32], Standard Error of Mean 2.462 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice
Statistical Analysis 2: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 12 hours of intra-oral exposure; Test type: Superiority; p = 0.2178, Mixed Models Analysis; Adjusted Mean Difference = 3.00, 95% CI 2-sided [-1.82 to 7.81], Standard Error of Mean 2.408 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice

10. Secondary Outcome: Adjusted Mean %RER at 4 and 12 Hours (Reference Dentifrice vs Placebo Control Dentifrice)
Description: as for outcome 2
Time Frame: as for outcome 7
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent RER
Arm/Group | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
percent RER
  At 4 hours of intra-oral exposure | -13.78 (3.022) | -48.89 (3.024)
  At 12 hours of intra-oral exposure | 0.19 (2.759) | -26.98 (2.760)
Statistical Analysis 1: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 4 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Adjusted Mean Difference = 35.12, 95% CI 2-sided [28.69 to 41.54], Standard Error of Mean 3.213 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice
Statistical Analysis 2: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 12 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Adjusted Mean Difference = 27.18, 95% CI 2-sided [21.14 to 33.21], Standard Error of Mean 3.018 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice

11. Secondary Outcome: Adjusted Mean EFU at 4 and 12 Hours (Reference Dentifrice vs Placebo Control Dentifrice)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: ITT population.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: microgram fluoride per square centimeter
Arm/Group | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
microgram fluoride per square centimeter
  At 4 hours of intra-oral exposure | 3.81 [3.42 to 4.25] | 2.20 [1.98 to 2.45]
  At 12 hours of intra-oral exposure | 3.89 [3.58 to 4.24] | 2.45 [2.25 to 2.66]
Statistical Analysis 1: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 4 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Geometric Mean Ratio = 1.73, 95% CI 2-sided [1.53 to 1.97]
Statistical Analysis 2: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 12 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Geometric Mean Ratio = 1.59, 95% CI 2-sided [1.42 to 1.78]

12. Secondary Outcome: Adjusted Mean ARR at 4 and 12 Hours (Reference Dentifrice vs Placebo Control Dentifrice)
Description: ARR was used to measure the resistance of the remineralized enamel to further acid softening. SMH technique was used to calculate ARR. Previously demineralized, sterilized bovine enamel specimens were placed intra orally using a palatal appliance. The enamel specimens were exposed to the dentifrice treatments in the mouth during the treatment application and allowed to remineralize intra orally under the action of the participant's saliva. The specimens were then removed from the palatal appliance and further treated with acid ex situ followed by additional SMH evaluations to yield ARR. The ARR was derived as 1 - [(E2-R)/(E1-B)] where: B = indentation length (μm) of sound enamel at baseline, E1 = indentation length (μm) after first erosive challenge (with a commercially available grapefruit juice), E2 = indentation length (μm) after second erosive challenge (with a commercially available grapefruit juice), R = indentation length (μm) after 4 and 12 hours in situ remineralization.
Time Frame: as for outcome 7
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
Number analyzed (Participants) | 33 | 33
ratio
  At 4 hours of intra-oral exposure | 0.580 (0.0214) | 0.273 (0.0214)
  At 12 hours of intra-oral exposure | 0.635 (0.0200) | 0.394 (0.0200)
Statistical Analysis 1: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 4 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Adjusted Mean Difference = 0.307, 95% CI 2-sided [0.252 to 0.362], Standard Error of Mean 0.0277 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice
Statistical Analysis 2: Comparison: Reference Dentifrice (Treatment C) vs Placebo Control Dentifrice (Treatment B); At 12 hours of intra-oral exposure; Test type: Superiority; p < .0001, Mixed Models Analysis; Adjusted Mean Difference = 0.242, 95% CI 2-sided [0.190 to 0.293], Standard Error of Mean 0.0257 — Adjusted mean difference was calculated as Reference Dentifrice minus Placebo Control Dentifrice

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 21 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product. A Serious Adverse Event (SAE) was a particular category of an AE where the adverse outcome is serious.
Arm/Group | Test Dentifrice (Treatment A) | Reference Dentifrice (Treatment C) | Placebo Control Dentifrice (Treatment B)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 4/33 | 1/33 | 5/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (Treatment A) (N=33) | Reference Dentifrice (Treatment C) (N=33) | Placebo Control Dentifrice (Treatment B) (N=33)
Pulpitis irreversible (Gastrointestinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Anxiety worsening (Psychiatric disorders) | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 1 | 0 | 0
Back Pain, Worsening (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT06242444/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT06242444/SAP_001.pdf